CLINICAL TRIAL: NCT05489991
Title: A Phase 1/2, Open-label, Multi-Center Study of Dually Armored Chimeric Antigen Receptor (CAR) T-cells (TmPSMA-02) in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: A Study of TmPSMA-02 Chimeric Antigen Receptor (CAR) T-cells in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was stopped Sponsor discretion. No patients were dosed.
Sponsor: Tceleron Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TmPSMA-0201
Record Dates: First submitted 2022-07-22; First posted 2022-08-05 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Chimeric Antigen Receptor (CAR); T-Cells; Prostate-Specific Membrane Antigen (PSMA); Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TmPSMA-02 (Experimental)
  Interventions: Biological: TmPSMA-02

INTERVENTIONS:
Biological: TmPSMA-02 — Intravenous administration of genetically modified autologous T-cells engineered to express a protein capable of recognizing the tumor antigen prostate-specific membrane antigen (PSMA) with a lentiviral vector to express anti-PSMA scFv, CD2 co-stimulatory domain and dually armored with a dominant negative TGFβ receptor and PD1.CD28 switch, will be infused intravenously on Day 0 as a single flat dose following standard lymphodepleting (LD) regimen.

SUMMARY:
An open-label, multi-center, Phase 1/2 study to determine the safety, tolerability, and feasibility of dosing adult patients with mCRPC with genetically modified autologous T-cells (TmPSMA-02) engineered to express a CAR capable of recognizing the tumor antigen prostate-specific membrane antigen (PSMA) and activating the T-cell.

DETAILED DESCRIPTION:
This is a Phase 1/2 single-arm study designed to identify the dose and regimen of TmPSMA-02 that can be safely administered intravenously following the lymphodepletion (LD) regimen to patients with mCRPC.

The Phase 1 dose escalation portion of the study will employ a Bayesian Optimal Interval (BOIN) Design to define the Maximum Tolerated Dose (MTD) and determine the Recommended Phase 2 Dose (RP2D). Dose-limiting toxicities (DLTs) will be assessed from the start of LD regimen through 28-days post infusion of TmPSMA-02.

The Phase 2 portion will employ a Simon's 2-stage design and include a single-arm of adult patients with mCRPC treated with the TmPSMA-02 at the RP2D.

It is anticipated that up to 30 patients will enroll in the Phase 1 portion of the study and up to 84 patients will enroll in the Phase 2 portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age.
* A confirmed histologic diagnosis of prostate cancer.
* Castrate levels of testosterone (< 50 ng/dL).
* Measurable disease (radiographic or Prostate Specific Antigen [PSA]) per PCWG3 criteria (see Appendix 3)
* Received at least 2 prior lines of systemic therapy for prostate cancer, including at least one second generation androgen receptor inhibitor (e.g., enzalutamide or apalutamide) or CYP17α inhibitor (e.g., abiraterone/ prednisone) and a taxane based regimen (e.g., docetaxel, cabazitaxel, etc). At least one line of prior therapy must be in the mCRPC setting. Note: Androgen deprivation therapy (ADT) with gonadotropin- releasing hormone (GnRH) agonist/antagonist does not count as a line of therapy nor does a first-generation nonsteroidal antiandrogen (e.g., bicalutamide, flutamide, etc.).
* Adequate vital organ function as defined by: (A) Estimated glomerular filtration rate (eGFR) eGFR ≥ 50 mL/min by Modification of Diet in Renal Disease criteria, (B) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x the upper limit of normal (ULN); patients with hepatic metastases ALT and AST ≤ 3.0 ULN. (C) Serum total bilirubin < 1.5 × ULN unless patient has known Gilbert's; if so, then serum bilirubin ≤ 3 mg/dL, or (D) Left ventricular ejection fraction ≥ 45%.
* Patients must have adequate hematologic reserve and must not be dependent on transfusions to maintain these hematologic parameters. Adequate hematologic reserve is defined as: (A) Hemoglobin ≥ 8 g/dL, (B) absolute neutrophil count ≥ 1000/ μL, or (C) Platelet count ≥ 75,000/μL.
* Patients who have not undergone bilateral orchiectomy must be able to continue GnRH therapy during the study.
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
* Toxicities from any previous therapy must have recovered to Grade 1 or to the baseline. Exceptions include non-clinically significant toxicities as a result of previous therapy (e.g., alopecia, hormonal changes, weight loss, etc).
* Patients of reproductive potential agree to use protocol-specified highly effective contraceptive methods

Exclusion Criteria:

* Active invasive cancer, other than the proposed cancer included in the study, within 2 years prior to screening. [Note: non-invasive cancers treated with curative intent (e.g., non-melanoma skin cancer may still be eligible], unless treated with curative intent, i.e., non-melanoma skin cancer.
* Prior treatment with autologous T-cell therapy. Note: Prior treatment with Sipuleucel-T is allowed.
* Patients who require chronic treatment with systemic corticosteroids (defined as a dose greater than the equivalent of prednisone 10 mg/day). Low-dose physiologic replacement therapy with corticosteroids equivalent to prednisone 10 mg/day or lower, topical steroids and inhaled steroids are acceptable.
* Prior allogeneic stem cell transplant.
* Active autoimmune disease (including, but not limited to, connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease or multiple sclerosis) or a history of severe autoimmune disease requiring prolonged immunosuppressive therapy. Patients should have stopped any immunosuppressive therapy within 6 weeks prior to Screening.
* Current infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV). Viral testing at Screening is required in all patients to rule out subclinical infections. Patients who are hepatitis B core antibody positive and hepatitis B surface antigen negative should have quantitative viral load measured. If viral load is undetectable, the patient may enroll and be monitored as per ASCO Guidelines.
* Seizure disorder requiring anti-epileptic medications.
* History of severe infusion reaction to monoclonal antibodies or biological therapies, or to study product excipients (e.g., human serum albumin, dimethyl sulfoxide [DMSO], dextran 40) that would preclude the patient safely receiving TmPSMA-02.
* History of or known predisposition to hemophagocytosis lymphohistiocytosis (HLH) or macrophage activation syndrome (MAS)
* Any active infection currently being treated with antibiotics, anti-virals or anti-fungal. Prophylactic anti-microbials are not exclusionary.
* Active or recent (within the past 6 months prior to leukapheresis) cardiovascular disease, defined as (1) New York Heart Association Class III or IV heart failure, (2) unstable angina or (3) a history of recent (within 6 months) myocardial infarction or sustained (> 30 second) ventricular tachyarrhythmias, (4) cerebrovascular accident.
* Active or uncontrolled medical or psychiatric condition that would preclude participation in the opinion of the Sponsor, Principal Investigator (PI) and/or their designee.
* Have inadequate venous access for or contraindications for the leukapheresis procedure. Central venous access is acceptable.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Phase 1: To evaluate the safety of TmPSMA-02 in adult patients with mCRPC | Up to 5 years
  Type, frequency, and severity of adverse events (AEs) and serious adverse events (SAEs)
Phase 1: To identify the recommended Phase 2 dose of TmPSMA-02 administered in combination with LD chemotherapy | Up to 5 years
  Frequency of DLTs and/or determination of the maximum tolerated dose (MTD)
Phase 2: To evaluate the objective response rate (ORR) per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 | Up to 5 years
  Objective Response Rate (ORR) by RECIST v1.1.

SECONDARY OUTCOMES:
Phase 1: To evaluate the preliminary antitumor activity of TmPSMA-02 according to RECIST v1.1 and the PCWG3 criteria | Up to 5 years
  Objective Response Rate (ORR), Duration of Response (DOR), PSA percent change from baseline at 12-weeks and maximal, change calculated at any timepoint Progression Free Survival (PFS) Radiographic progression free survival (rPFS) Overall Survival (OS)
Phase 1: To assess the clinical and manufacturing feasibility of TmPSMA-02 | Up to 5 years
  Clinical: proportion of patients enrolled on this protocol who do not receive TmPSMA-02 cells for any reasons not related to manufacturing (see below) Manufacturing: Proportion of patients whose leukapheresis product results in manufacturing failure for any reason
Phase 2: To evaluate the safety and tolerability of TmPSMA-02 in adult patients with mCRPC | Up to 5 years
  Type, frequency, severity of AEs, SAEs
Phase 2: Evaluate the anti-tumor activity of TmPSMA-02 according to Prostate Cancer Working Group 3 (PCWG3). | Up to 5 years
  Duration of Response (DOR), PSA percent change from baseline at 12-weeks and maximal change calculated at any timepoint, Progression Free Survival (PFS), Radiographic progression free survival (rPFS), Overall Survival (OS)
Phase 2: Describe pharmacokinetic factors of TmPSMA-02 in peripheral blood | Up to 5 years
  Expansion and persistence of CAR T-cells by molecular detection of CAR-specific sequences in peripheral blood
Phase 2: Evaluate changes in patient reported health-related outcomes following treatment with TmPSMA-02 | Up to 5 years
  Evaluate changes in health-related outcomes following treatment with TmPSMA-02 using the Functional Assessment of Cancer Therapy - Prostate Cancer (FACT-P)

CONTACTS AND LOCATIONS:
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States